CLINICAL TRIAL: NCT02810236
Title: Focal Breast Pain: Does a Normal Ultrasound Provide Reassurance?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00070445
Record Dates: First submitted 2016-05-23; First posted 2016-06-22 (Estimated); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Breast Diseases; Mastodynia; Anxiety
Keywords: Focal breast pain; Directed Ultrasound; Reassurance; Anxiety
MeSH Terms: conditions — Breast Diseases; Mastodynia; Anxiety Disorders | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No ultrasound (Active Comparator): No ultrasound recommended. Discussion with radiologist.
  Interventions: Behavioral: Discussion
- Ultrasound (Active Comparator): Ultrasound recommended.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound will be performed.
  Arms: Ultrasound
Behavioral: Discussion — Radiologist will discuss with the patient the findings on mammogram.
  Arms: No ultrasound

SUMMARY:
The investigator hypothesizes that a benign directed ultrasound, when performed after a normal digital mammogram, will provide women with focal breast pain additional reassurance that the etiology of their symptom is benign. 160 women over the age of thirty with focal breast pain who present to the Breast Imaging Clinic for evaluation between 3/1/2016 - 7/1/2018 will be selected and randomized to three groups using a block randomization technique. All study participants will complete a survey assessing psychosocial factors, then receive a digital mammogram. Patients with a negative mammogram will continue on with the study and will either have a conversation about their negative mammogram with a radiologist or receive a directed ultrasound. A second survey will be conducted assessing psychosocial factors. All study participants who did not receive an ultrasound will receive an ultrasound so that all study participants are provided with the standard of care for focal breast pain. The results of the survey will be compared and appropriate statistical analyses such as an Analysis of Variance (ANOVA) test will be conducted to determine any statistically significant differences between the three randomized groups. The risks/safety issues of this study are believed to be minimal.

DETAILED DESCRIPTION:
Protocol Title: Focal Breast Pain: Does a normal ultrasound provide reassurance?

Purpose of the Study: The investigator hypothesizes that a benign directed ultrasound, when performed after a normal digital mammogram, will provide women with focal breast pain additional reassurance that the etiology of their symptom is benign.

Background & Significance: Breast pain is one of the most common symptoms for which women seek medical care. While up to 80% of women experience breast pain at some point in their lives, most commonly breast pain results from a benign etiology such as trauma, infection, pregnancy, lactation, or simple cysts. In contrast, breast cancer is only reported in up to 7% of women presenting with focal breast pain. Despite the uncommon association between breast cancer and focal breast pain, a diagnostic imaging workup is often requested. Current American College of Radiology (ACR) Appropriateness Criteria guidelines rate the use of mammography and ultrasound for the evaluation of non-cyclical, focal, unilateral or bilateral breast pain in patients 30 years and older as "may be appropriate." Traditionally both mammography and ultrasound are performed in women over the age of 30, who present with noncyclical, focal breast pain as imaging can often exclude a treatable benign cause of pain and/or provide reassurance.

The investigator recently completed a retrospective study evaluating the utility of digital mammography and directed ultrasound in women with focal breast pain. It was observed that performing directed ultrasound following digital mammography was potentially beneficial in women with mammographically dense breast tissue. In contrast, the investigator demonstrated that directed ultrasound in conjunction with digital mammography was of low utility in women with non-dense breast tissue. These findings suggest that directed ultrasound might be unnecessary in the work up of focal breast pain for women with non-dense breast tissue.

However, there is anecdotal evidence that a directed ultrasound yielding benign findings following a normal digital mammogram might further reassure women that the cause of focal breast pain is benign. These potential psychological benefits may drive the continued use of ultrasound in the work up of focal breast pain, even though their diagnostic utility is low.

Design and Procedures:

Subject Selection, Recruitment, and Compensation

The study team (Principal investigator (PI), Co-PI, and Study coordinator) will select up to 160 women, who present to the Breast Imaging Clinic for evaluation of focal breast pain between 3/1/2016 - 7/1/2018. Inclusion criteria include women over the age of 30 with primary focal breast pain, i.e. pain localizable by the patient to within one breast quadrant without other associated symptoms. Women with diffuse, radiating, or axillary pain, associated palpable findings at the site of pain, skin changes (erythema, thickening) or nipple changes (discharge, retraction), currently pregnant or breast-feeding, history of recent trauma or infection of the affected breast, and history of ipsilateral breast cancer will be excluded.

Based on the investigator's clinical judgement, the investigator anticipates a minimum effect size of d=.4 for anxiety. A sample size of n =80 per group (total n = 160) has power of 0.8 to detect differences with an effect size of d=.4 using a one-tailed alpha = .05.

Study participants will include women referred for imaging because of focal breast pain and women who report focal breast pain to the technologist or radiologist prior to imaging. Once a patient is identified as a possible candidate, the PI, Co-PI, or study coordinator will look at electronic medical record, Epic. to see if they meet inclusion criteria and do not have any exclusion criteria. If there are none, the patient will be approached to see if they are willing to participate in the study. While the number of patients who present in a typical week to Duke with focal breast pain has not been studied, anecdotally, approximately 1-2 patients per day have been evaluated for focal breast pain. Study participants will not be compensated.

Consent Process

Study participants will include women referred for imaging because of focal breast pain and women who report focal breast pain to the technologist or radiologist prior to imaging. Once a patient is identified as a possible candidate, the PI, Co-PI, or study coordinator will look at Epic to see if they meet inclusion criteria and do not have any exclusion criteria. If there are none, the patient will be approached to see if they are willing to participate in the study. Only a member of the study team (Karen Johnson, MD, Lars Grimm, MD, and Michael Cho, MD) will approach a potential participant for the consent process. If a member of the study team is not available, the potential subject will not be recruited. Subjects who are able to provide legally effective consent will be recruited.

While the number of patients who present in a typical week to Duke with focal breast pain has not been studied, anecdotally, approximately 1-2 patients per day have been evaluated for focal breast pain.

This study will serve as the 3/2 research project for Michael Cho, MD. Dr. Cho has requested 37 weeks of dedicated research time during his 4th year to recruit patients. Dr. Cho will continue to recruit patients during his Breast imaging fellowship if needed. As such, Dr. Cho will be primarily responsible for the consent process. Dr. Cho will work with Steve Shipes to learn about the consent process and Maestro data entry.

Study Design

Once a patient volunteers to participate, the investigator will utilize a block randomization technique to randomize the study participants into two groups (Group A and B), ensuring comparable numbers across the study groups. The patient will then be consented. Pertinent demographic and medical data will also be collected.

All included study participants will be asked to complete a short survey, based on the State Anxiety scale of the State-Trait Anxiety Inventory (STAI) (18). This survey will primarily assess psychosocial metrics, including, but not limited to anxiety, comfort, and level of concern for malignancy.

All study participants will receive a digital mammogram, which is the standard of care for patients presenting with focal breast pain. Patients with no imaging correlate to the focal breast pain (Breast imaging-reporting and data system (BI-RADS) 1 and 2) will continue on with the study. Patients with an imaging finding at the site of focal pain (BI-RADS 0, 4, or 5) will be excluded from the study and receive the standard care that is appropriate for the imaging finding.

Women with BI-RADS 1 and 2 digital mammograms will proceed with the study and be informed of their imaging findings. Study participants randomized to Group A will receive their mammogram results from a Breast imaging fellow or fellowship trained Breast imaging radiologist. Participants in Group B will receive their mammogram results from a Breast imaging fellow or fellowship trained Breast imaging radiologist and additionally receive a directed ultrasound in the area of focal pain, which is the standard of care for focal breast pain.

All study participants will be asked to complete a second survey, based on the State Anxiety scale of the State-Trait Anxiety Inventory.

Participants in Groups A will receive a directed ultrasound of their breast at the end of the visit ensuring that all women receive the standard of care. One of the research collaborators will approach subjects in groups A following the 2nd survey to disclose the minor deception and explain to the subjects the necessity of the deception for the purposes of the study. The collaborator will also explain that the current standard of care for patients with focal breast pain is a targeted ultrasound. The standard of care ultrasound will then be performed by a Breast imaging fellow or fellowship trained breast radiologist.

Risk/Benefit Assessment

The risks of this study are believed to be minimal, including the potential loss of confidentiality. The digital mammogram and directed ultrasound patients will receive are the standard of practice for women with focal breast pain. Women in this study would have received these imaging tests regardless of their participation in the study and therefore the potential risks of imaging are not considered additional risks of this study.

Costs to the Subject: There are no projected direct financial costs to the subjects involved in this study.

Data Analysis & Statistical Considerations: The results of the survey will be compared and appropriate statistical analyses including but not limited to analysis of variance and multiple two sample t-tests conducted to determine any statistically significant differences between the three randomized groups.

Data & Safety Monitoring: There are no anticipated safety concerns. The study coordinator (MC) will be responsible for the data collection and storage. Paper surveys will be stored in a locked cabinet in the Breast imaging reading room (Cancer Center Room 2S33) in the Cancer Center Breast Imaging Department (Clinic 2-1) which is accessible by badge only. Any digital data will be stored on an encrypted external hard drive (Western Digital) with a backup on Duke approved cloud storage (Box) and DTHS managed shared drive.

Privacy, Data Storage & Confidentiality: A de-identification code will be assigned to the patients to be used as their identifier. The linking code identifying the subject will be kept for the duration of the study and will be securely stored on an encrypted external hard drive (Western Digital) with a backup on Duke approved cloud storage (Box) and DTHS managed shared drive.

ELIGIBILITY:
Inclusion Criteria:

* women
* over the age of 30
* primary focal breast pain, i.e. pain localizable by the patient to within one breast quadrant without other associated symptoms.

Exclusion Criteria:

* diffuse, radiating, or axillary pain
* associated palpable findings at the site of pain
* skin changes (erythema, thickening)
* nipple changes (discharge, retraction)
* currently pregnant or breast-feeding
* history of recent trauma or infection of the affected breast
* history of ipsilateral breast cancer will be excluded.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change in anxiety using modified STAI questionnaire | baseline, day 1
  Measure change in anxiety following intervention using modified STAI

CONTACTS AND LOCATIONS:
Overall Officials: Michael Taylor-Cho, MD, Principal Investigator — Duke University; Lars Grimm, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masroor I, Afzal S, Sakhawat S, Khan N, Beg MA, Kawal D. Negative predictive value of mammography and sonography in mastalgia with negative physical findings. J Pak Med Assoc. 2009 Sep;59(9):598-601. PMID 19750852
- [Background] Mansel RE. ABC of breast diseases. Breast pain. BMJ. 1994 Oct 1;309(6958):866-8. doi: 10.1136/bmj.309.6958.866. No abstract available. PMID 7950621
- [Background] Howard MB, Battaglia T, Prout M, Freund K. The effect of imaging on the clinical management of breast pain. J Gen Intern Med. 2012 Jul;27(7):817-24. doi: 10.1007/s11606-011-1982-4. Epub 2012 Jan 31. PMID 22331398
- [Background] Morrow M. The evaluation of common breast problems. Am Fam Physician. 2000 Apr 15;61(8):2371-8, 2385. PMID 10794579
- [Background] Jokich P, Newell MS, Bailey L, et al. ACR Appropriateness Criteria® breast pain. Available at http://www.acr.org/~/media/ACR/Documents/AppCriteria/Diagnostic/ BreastPain.pdf. American College of Radiology. Accessed June 20, 2015.
- [Background] Barton MB, Elmore JG, Fletcher SW. Breast symptoms among women enrolled in a health maintenance organization: frequency, evaluation, and outcome. Ann Intern Med. 1999 Apr 20;130(8):651-7. doi: 10.7326/0003-4819-130-8-199904200-00005. PMID 10215561
- [Background] Preece PE, Mansel RE, Bolton PM, Hughes LM, Baum M, Gravelle IH. Clinical syndromes of mastalgia. Lancet. 1976 Sep 25;2(7987):670-3. doi: 10.1016/s0140-6736(76)92477-6. PMID 60528
- [Background] Srivastava A, Mansel RE, Arvind N, Prasad K, Dhar A, Chabra A. Evidence-based management of Mastalgia: a meta-analysis of randomised trials. Breast. 2007 Oct;16(5):503-12. doi: 10.1016/j.breast.2007.03.003. Epub 2007 May 16. PMID 17509880
- [Background] Harvey JA, Mahoney MC, Newell MS, Bailey L, Barke LD, D'Orsi C, Hayes MK, Jokich PM, Lee SJ, Lehman CD, Mainiero MB, Mankoff DA, Patel SB, Reynolds HE, Sutherland ML, Haffty BG. ACR appropriateness criteria palpable breast masses. J Am Coll Radiol. 2013 Oct;10(10):742-9.e1-3. doi: 10.1016/j.jacr.2013.06.013. PMID 24091044
- [Background] Vaidyanathan L, Barnard K, Elnicki DM. Benign breast disease: when to treat, when to reassure, when to refer. Cleve Clin J Med. 2002 May;69(5):425-32. doi: 10.3949/ccjm.69.5.425. PMID 12022387
- [Background] Noroozian M, Stein LF, Gaetke-Udager K, Helvie MA. Long-term clinical outcomes in women with breast pain in the absence of additional clinical findings: mammography remains indicated. Breast Cancer Res Treat. 2015 Jan;149(2):417-24. doi: 10.1007/s10549-014-3257-3. Epub 2015 Jan 6. PMID 25556516
- [Background] Olcucuoglu E, Yilmaz G. Mastodynia: is imaging necessary in young patients? Ulus Cerrahi Derg. 2013 Mar 1;29(1):17-9. doi: 10.5152/UCD.2013.04. eCollection 2013. PMID 25931836
- [Background] Tumyan L, Hoyt AC, Bassett LW. Negative predictive value of sonography and mammography in patients with focal breast pain. Breast J. 2005 Sep-Oct;11(5):333-7. doi: 10.1111/j.1075-122X.2005.00018.x. PMID 16174154
- [Background] Leddy R, Irshad A, Zerwas E, Mayes N, Armeson K, Abid M, Cluver A, Campbell A, Ackerman S, Lewis M. Role of breast ultrasound and mammography in evaluating patients presenting with focal breast pain in the absence of a palpable lump. Breast J. 2013 Nov-Dec;19(6):582-9. doi: 10.1111/tbj.12178. Epub 2013 Sep 9. PMID 24011215
- [Background] Leung JW, Kornguth PJ, Gotway MB. Utility of targeted sonography in the evaluation of focal breast pain. J Ultrasound Med. 2002 May;21(5):521-6; quiz 528-9. doi: 10.7863/jum.2002.21.5.521. PMID 12008815
- [Background] Duijm LE, Guit GL, Hendriks JH, Zaat JO, Mali WP. Value of breast imaging in women with painful breasts: observational follow up study. BMJ. 1998 Nov 28;317(7171):1492-5. doi: 10.1136/bmj.317.7171.1492. PMID 9831579
- [Background] Preece PE, Mansel RE, Hughes LE. Mastalgia: psychoneurosis or organic disease? Br Med J. 1978 Jan 7;1(6104):29-30. doi: 10.1136/bmj.1.6104.29. PMID 620138
- [Background] Spielberger CD. Manual for the State-Trait Anxiety Inventory (Form Y). Palo Alto, CA: Mind Garden; 1983.